CLINICAL TRIAL: NCT03515642
Title: Effect of Two Exercise Programme on Gut Microbiota, Hepatic Metabolism and Adipokines in Sedentary Adults With Overweight
Brief Title: Exercise, Gut Microbiota in Sedentary Adults With Overweight
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant due to PI not employment at University.
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Universidad de Santiago de Chile (Other); Universidad Pública de Navarra (Other); Universidad del Rosario (Other); NavarraBiomed Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DVO005-1-338-CEI882
Record Dates: First submitted 2018-04-21; First posted 2018-05-03 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Metabolic Disturbance
Keywords: Gut microbiota; Hepatic function; Obesity; Exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT group (Experimental): The HIIT modality consisted of 30-40 minutes (min) of steady-state, high-intensity training 3 d/wk on a stationary bicycle at the target heart rate (HR) range equivalent to 85% to 95% of the individual's maximum oxygen consumption rate (VO2max). Exercise will be performed at three sessions per week. All sessions will be supervised by an exercise physiologist during 6-weeks.
  Interventions: Behavioral: HIIT group
- SIT group (Active Comparator): The SIT modality consisted of 6 to 10 repetitions of a 30 s segment of all-out exercise interspersed with 2 min of recovery, 3 d/wk on a stationary bicycle at the target heart rate (HR) range equivalent to 90% to 95% of the individual's maximum oxygen consumption rate (VO2max).
  Interventions: Behavioral: HIIT group

INTERVENTIONS:
Behavioral: HIIT group — Physical Training
  Other Names: High/low volume exercise

SUMMARY:
This project offers the opportunity to obtain detailed measurements on the health of body composition, metabolic health, and intestinal microbial diversity in overweight adults; moreover to provide information about the effects of physical exercise on them. The aim of the research is to advance in the understanding of the mechanisms induced by physical exercise, which includes the measurement of nutritional parameters, clinical and biochemical biomarkers of hepatic/cardiometabolic health, as well as the application of differential proteomics technologies by means of Arrays of cytokines and intestinal microbiome, making this study a novel and pioneer in sensitive areas of primary health care in Latin America.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Sedentary males
* BMI>25 kg/m2, on a stable body weight for the last 3 months

Exclusion Criteria:

* Acute or chronic illness
* Use of antibiotics the past 2 months
* Smoking

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline in the gut microbiota composition measured by amplicon sequencing
Plasma metabolomic profile | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline in the metabolomic profile will be also evaluated by a HPLC-MS approach

SECONDARY OUTCOMES:
Plasma hepatokines | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline in the Chemerin will be measured using ELISA kits
Plasma hepatokines | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline in the Selenoprotein P will be measured using ELISA kits
Plasma hepatokines | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline in the Fetuin-A will be measured using ELISA kits
Plasma hepatokines | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline in the FGF21 (fibroblast growth factor 21) Leukocyte cell-derived will be measured using ELISA kits
Glucose | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline will be also evaluated by a spectroscopy
Insulin | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline will be also evaluated by a ELISA
Glycated hemoglobin | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline will be also evaluated by a ELISA
Bioinflammatory blood markers | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline measure of plasma IL-1 concentrations measured ELISA
Bioinflammatory blood markers | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline measure of plasma IL6 concentrations measured ELISA
Bioinflammatory blood markers | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline measure of plasma TNF-alfa concentrations measured ELISA
Bioinflammatory blood markers | Baseline, and 6 weeks immediately after the interventions ends
  Change from Baseline measure of plasma CRP concentrations measured ELISA
Body composition | Baseline, and 6 weeks immediately after the interventions ends
  Differences in body weight (kilograms) measured by DXA
Body composition | Baseline, and 6 weeks immediately after the interventions ends
  Differences in body fat (%) measured by DXA
Body composition | Baseline, and 6 weeks immediately after the interventions ends
  Differences in mass muscle measured by DXA
Physical fitness | Baseline, and 6 weeks immediately after the interventions ends
  Differences in Muscular strength (handgrip test) in kg
Physical fitness | Baseline, and 6 weeks immediately after the interventions ends
  Differences in Maximum Oxygen Consumption (VO2 max K5 Gas Analyser) in ml/kg/min
Energy substrate oxidation | Baseline, and 6 weeks immediately after the interventions ends
  Fat and carbohydrate oxidation in the fasted and postprandial state measured before and after the interventions using indirect calorimetry (K5 cosmed)
Resting Metabolic Rate | Baseline, and 6 weeks immediately after the interventions ends
  Resting metabolic rate was measured before and after the interventions (K5 Cosmed)

CONTACTS AND LOCATIONS:
Locations (1):
- Robinson Ramírez-Vélez, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No